CLINICAL TRIAL: NCT00922506
Title: Comparison of the Efficacy and Safety of Combination Treatment With Doxazosin Plus TolterodineSR 2 mg vs Doxazosin Plus TolterodineSR 4 mg in Men With an OAB/BPO: Randomized Controlled Study"
Brief Title: Combination Treatment With Doxazosin Plus TolterodineSR 2 mg Versus 4mg in Men With an Overactive Bladder (OAB) and Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor,MD,PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-08-092
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Overactive Bladder; Benign Prostatic Hyperplasia
Keywords: Overactive bladder; Benign prostate hyperplasia; Doxazosin; Tolterodine
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- doxazosin plus tolterodine SR 2 mg (Experimental): doxazosin plus tolterodine SR(2 mg, qd) for 12 weeks
  Interventions: Drug: doxazosin plus tolterodine SR
- doxazosin plus tolterodine SR 4 mg (Experimental): doxazosin plus tolterodine SR(4 mg,qd) for 12 weeks
  Interventions: Drug: doxazosin plus tolterodine SR

INTERVENTIONS:
Drug: doxazosin plus tolterodine SR — doxazosin plus tolterodine SR(2 mg, qd)for 12 weeks or (4 mg, qd) for 12 weeks
  Other Names: Cadura XL 4mg or 8mg; Detrusitol SR 2mg

SUMMARY:
OAB occurs in approximately 50% to 75% of men with BPO and up to 38% of men with BPO continue to suffer from OAB after relief the obstruction.Symptoms of OAB are more bothersome than the voiding complaints of slow stream and hesitancy. However, the patients with both BPO and OAB are often not treated with muscarinic receptor antagonists due to concern that they will experience acute urinary retention.

Tolterodine is a potent and pure muscarinic receptor antagonist that was developed specifically for the treatment of overactive bladder. Recently, studies revealed that tolterodine was effective, safe and well tolerated in adults with OAB and urodynamically confirmed BPO.However, the optimal dosage of antimuscarinic for the treatment of OAB coexisting BPO was not yet fully assessed. In real clinical situation, some patients complain voiding difficulty after addition of antimuscarinics and want to stop antimuscarinics.It is probable that a lower dosage of antimuscarinics combined with alpha-adrenergic antagonists can be used safely in OAB patients with BOO, with the same efficacy.

This study is designed to investigate the optimal doses of tolterodine SR in combination with doxazosin in men with both BOO and OAB based on efficacy, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 50 ≤ and ≤ 80 years
* Proven bladder outlet obstruction (BOO, Abrams/Griffith score >20) on urodynamic study
* Symptoms of OAB as verified by the 3 day voiding diary, defined by:

  1. symptoms of urinary urgency (defined as a level of ≥3 in a 5 point urgency scale) at least two episode per 24 hours and
  2. symptoms of urinary frequency (8 micturitions per 24 hours)
* Total International Prostate Symptom Score (IPSS) of 12 or higher
* IPSS quality-of-life (QOL) item score of 3 or higher
* A rating of the bladder condition at Baseline prior to randomization as "Some Moderate Problems", "Severe Problems", or "Many Severe Problems" on the Patient Perception of Bladder Condition (PPBC) questionnaire.
* Ability and willingness to correctly complete the micturition diary and questionnaire
* Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

* Patients have a baseline post-void residual (PVR) which exceeded 150 mL.
* Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention.
* Symptomatic acute urinary tract infection (UTI) during the screening period.
* Treatment within the 14 days preceding randomization, or expected to initiate treatment during the study with any anticholinergic drugs and drug treatment for overactive bladder.
* A 5-alpha reductase inhibitor if started less than 3 months prior to screening.
* Patients with previous urethral, prostate or bladder neck surgery.
* Patients with cancer of any type including cancer of the prostate or bladder, uncontrolled medical condition including psychiatric disease or life threatening illness.
* Patients with Parkinson's disease, stroke, multiple sclerosis, spinal cord disease.
* Patients with suspected neurogenic bladder disorder.
* Patients with urethral stricture or bladder neck contracture.
* Serum PSA 4ng/ml (only patients with no malignancy by prostate biopsy can be included).

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Numeric change of urgency episodes per 24 hours | 12 weeks of treatment

SECONDARY OUTCOMES:
Changes in voiding diary parameters | 12 weeks of treatment
Change in symptom questionnaires | 12 weeks
Patient-Rated Global Assessments of Treatment Benefit, Satisfaction, and Willingness to Continue | 12 weeks
Change of uroflowmetry and PVR | 12 weeks
Incidence of acute urinary retention | during all study periods

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401